CLINICAL TRIAL: NCT04254952
Title: The Validity and Reliability of the Turkish Version of the Nijmegen Questionnaire in Evaluating Respiratory Dysfunction in Asthmatic Patients
Brief Title: Turkish Version of Nijmegen Questionnaire
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aslihan Cakmak, Research Assistant, Hacettepe University
Other Study IDs: GO 20/199
Record Dates: First submitted 2019-10-15; First posted 2020-02-05 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Hyperventilation Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to provide Turkish version of Nijmegen Questionnaire for the evaluation of respiratory dysfunction in asthmatic subjects. The incidence of hyperventilation syndrome in asthmatic patients can be determined with the results of the study.

DETAILED DESCRIPTION:
Nijmegen Questionnaire allows to assess and identify respiratory symptoms and dysfunction, and to assess unexplained respiratory symptoms and symptoms of hyperventilation syndrome. Determining whether Turkish version of Nijmegen Questionnaire is a valid and reliable tool in asthmatic individuals will guide researchers for further studies on identifying appropriate treatment approaches for the patient and developing different treatment strategies. Hyperventilation syndrome is a recognized form of respiratory dysfunction associated with biochemical factors. Hyperventilation syndrome is defined as breathing above the body's metabolic requirements. This results in decreased carbon dioxide pressure in the arterial blood, respiratory alkalosis, and increased symptoms. Complex symptoms such as shortness of breath, chest tightness, paresthesia, anxiety, and dizziness may occur. There is no laboratory test which is the gold standard in the diagnosis of hyperventilation syndrome. If it is concluded that the Turkish version of the Nijmegen Questionnaire is a valid and reliable test in individuals with asthma, a new tool will be introduced to the literature for the evaluation of pulmonary dysfunction in asthmatic individuals.

ELIGIBILITY:
Inclusion Criteria:

* Having mild to moderate clinically stable asthmatic patients
* Being able to cooperate
* Being 18 years old or older

Exclusion Criteria:

* Having severe orthopedic, neurological, cardiovascular disorders or cognitive problems
* Unable to cooperte

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Asthmatic patients
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2021-02-21 (Actual); Study Completion 2021-02-21 (Actual)

PRIMARY OUTCOMES:
Dyspnea perception | 1st day
  Dyspnea will be evaluated with a modified Borg scale. The modified Borg scale is a category scale that evaluates dyspnea between the scores of 0-10. Patients will be asked to mark the appropriate value on the scale.
Breathe-holding time | 1st day
  Individuals are asked to hold their breaths in the sitting position by closing their nostrils and in functional residual volume (after a normal exhalation). In order to eliminate the learning effect, the measurement is repeated three times and the averages of the times are recorded in seconds.
End-tidal CO2 measurement | 1st day
  A portable capnograph with a nasal cannula will be used for the measurement of mean ETCO2 and resting respiration rate over a ten-minute period. Individuals will be asked to breathe through the nose and not speak during the measurement.
Asthma control test | 1st day
  Test is used to evaluate asthma control. The questionnaire consists of five items. The total test score ranges from 5 (weak control) to 25 (fully controlled) (14). A total score of <20 indicates uncontrollable asthma.
Nijmegen Questionnaire | 1st day
  The Nijmegen Questionnaire has been validated as a screening tool for the detection of hyperventilation syndrome (HVS), consisting 16 items. A score of over 23 out of 64 suggests a positive diagnosis of HVS. It has also been used to detect dysfunctional breathing in patients with asthma.

SECONDARY OUTCOMES:
Quality of life questionnaire | 1st day
  The overall quality of life will be determined by the Nottingham Health Profile (NHP). The NHP consists of 38 substances that the individual can complete without the need for a person. The questionnaire has six sub scales: energy (3 items), pain (8 items), emotional reactions (9 items), sleep (5 items), social isolation (5 items) and physical mobility (8 items). For each subsection there is a possible range of points ranging from 0-100 points. Higher scores indicate more limitations in quality of life.
Disease-specific quality of life | 1st day
  Disease-specific quality of life will be determined by the Asthma Quality of Life Questionnaire (AQLQ). The Asthma Quality of Life Questionnaire was found to be valid and reliable in Turkish. The quality of life questionnaire in individuals with asthma is a 32-item disease-specific questionnaire in four health domains, including activity limitation (11 items), symptoms (12 items), emotional function (5 items), and environmental stimuli (4 items). Scores range 1-7, with higher scores indicating better quality of life.
Assessment of anxiety and depression | 1st day
  The Beck Depression Inventory (BDI) measures physical, emotional, cognitive, and motivational symptoms of depression. The aim of the scale is to determine the level of depression symptoms and the change in severity. BDI is a scale that includes 21 self-assessment sentences and there are four options in each symptom category. Each item is scored between 0-3 points and the total score varies between 0 and 63. The validity and reliability study of the scale was conducted in Turkish. The cut-off value of the Turkish form was determined to be 17.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Inal-Ince, Prof, Study Director — Hacettepe University; Gul Karakaya, Prof, Principal Investigator — Hacettepe University; Aslihan Cakmak, MSc, Principal Investigator — Hacettepe University; Senem Simsek, MSc, Principal Investigator — Hacettepe University
Locations (1):
- Aslihan Cakmak, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No